CLINICAL TRIAL: NCT05067621
Title: Semaglutide, 2.4mg, Once Weekly: Effects on Beta-cell Preservation and Reduction of Intrahepatic Triglyceride Content in Obese Youth With Prediabetes (IGT)/Early Type 2 Diabetes (T2D) and Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Semaglutide Effects in Obese Youth With Prediabetes/New Onset Type 2 Diabetes and Non-Alcoholic Fatty Liver Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Caprio, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000031181; 2R01DK111038-06A1 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-10-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus; Impaired Glucose Tolerance; Non-Alcoholic Fatty Liver Disease; Obesity, Childhood
Keywords: Prediabetes; NAFLD; Impaired Glucose Tolerance; Semaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Non-alcoholic Fatty Liver Disease; Pediatric Obesity; Prediabetic State | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Participants will undergo baseline tests at the beginning of the study and will be randomized to receive experimental drug or placebo. Dose escalation will be achieved within 16 weeks to reach up to 2.4mg of Semaglutide, weekly, which they will be on for 6 months. All tests will be repeated after 6 months of treatment followed by a wash-out period of 3 months, after which the same tests will be repeated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Yale Investigational Drug Services Pharmacy will handle the masking of drug and placebo pens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receive treatment (Experimental): Semaglutide (Wegovy) pen is a subcutaneous injection
  Interventions: Drug: Semaglutide Pen Injector
- Placebo (Placebo Comparator): The placebo pen is almost exactly the same as the Wegovy subcutaneous injection except it does not contain the active ingredient, Semaglutide.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Semaglutide (Wegovy) pen is a subcutaneous injection that contains 2.4mg/0.75mL of active ingredient. The injection pen can deliver doses of 0.24mg, 0.5mg, 1.0mg, 1.7mg, and 2.4mg.
  Other Names: Wegovy
  Arms: Receive treatment
Drug: Placebo — Injection pen contains excipients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand the role of GLP-1 in the pathogenesis of T2D in youth and explore their potential salutary effects and ability to delay the progressive loss of ß-cell function and reduce hepatic steatosis in youth with prediabetes/new onset T2D and NAFLD.

DETAILED DESCRIPTION:
In a recent publication by the TODAY Group Study, it was reported that "diabetes-related complications appear early in youth-onset T2D and accumulate rapidly at a mean age of 26.4 years," and 60.1% of participants developed at least one microvascular complication. The same has been reported in RISE Studies and was suggested that the rapid decline in β-cell function and its insensitivity to two of the most frequently used treatments for T2D in pediatrics is further aggravated by the rising prevalence in NAFLD. These alarming results indicate a pressing need for effective and innovative approaches at preserving β-cell function and reducing hepatic steatosis in obese youth in order to prevent disease progression and associated complications.

This study will provide mechanistic insights in support of a GLP-1 analog, Semaglutide, 2.4 mg weekly, therapy for prediabetes, new onset T2D and NAFLD in youth. The study design is a randomized, double-blind, placebo-controlled, clinical trial (RCT) using Semaglutie (Wegovy up to 2.4mg) for 6 months followed by a wash-out period of 3 months.

ELIGIBILITY:
Inclusion Criteria

* Subjects diagnosed with Pre-impaired glucose tolerance (pre-IGT) (2h glucose ≥ 130 mg/dl to ≤ 200 mg/dl post-OGTT) OR impaired glucose tolerance (2h glucose ≥140 to <200 mg/dl post-OGTT OR HbA1c ≥5.7% to <6.5%), OR new-onset T2D (≤24 months duration, 2h glucose >200 and HbA1c >6.5% to10%) treated with stable metformin dose (stable metformin dose is defined as at least 1000 mg daily or the maximum tolerated dose for 12 months or less)
* PDFF of ≥ 8%
* Male or female, aged 10 to <21 years at the day of randomization, in puberty (pubertal stage will be assessed by pediatric Endocrinologists Dr. Samuels and Dr. Hu) (girls and boys: Tanner stage II-IV); girls who begin menstruating must have a negative pregnancy test during the study
* Weight ≥ 54kg
* BMI ≥ 85% but ≤ 40 kg/m2
* Good general health (normal kidney function, amylase, and lipase levels)
* Informed consent from a legally acceptable representative (LAR) and child assent from the subject obtained before any trial-related activities (trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial)
* Ability and willingness to adhere to the protocol including self-measurement of plasma glucose according to the protocol.

Exclusion Criteria

* Known or suspected hypersensitivity to trial product(s) or related products.
* Receipt of any investigational medicinal product within 30 days before screening.
* Prepubertal participants (Tanner stage 1)
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive methods.
* Having a diagnosis of:

  * Type 1 diabetes o Maturity onset diabetes of the young (MODY) o History or presence of Pancreatitis (acute or chronic) o Presence of endocrinopathies (e.g., Cushing syndrome) o Cardiac, renal or pulmonary or other chronic illness o Known history of heart disease (including history of clinically significant arrhythmias or conduction delays on ECG, or new clinically significant arrhythmias or conduction delays on ECG identified at visit 1) o Family or personal history of MEN type 2 or medullary thyroid carcinoma (family is defined as a first-degree relative)o Any other disorder which, in the opinion of the investigator, might jeopardize subject's safety or compliance with the protocol
* Any laboratory safety parameter at screening outside the below extended laboratory ranges: o Baseline creatinine >1.0mg o Hypertriglyceridemia)(>500 mg/dl)

  * Calcitonin equal or above 50 ng/L at screening o Body Mass Index (BMI) ≤ 25.0 at the screening visit o ALT ≥5 times the upper normal limit (UNL) o Creatinine >UNL for age in children unless renal function is proven normal by further assessments at the discretion of the investigator
* Known hypoglycemic unawareness.
* Recurrent severe hypoglycemic episodes within the last year as judged by the investigator.
* Uncontrolled hypertension treated or untreated >99th percentile for age and gender in children and adolescents.
* Treatment with any medication for the indication of diabetes other than stated in the inclusion criteria in a period of 90 days before screening.
* Taking medication, based on the investigator's judgement, that may cause significant weight gain or loss (e.g., antipsychotic, steroid, anti-obesity medication).
* Presence or history of malignant neoplasm within 5 years prior to the day of screening.Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.
* Positive insulinoma associated-protein 2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies.

Mental health:

* History of major depressive disorder within 2 years before screening
* Diagnosis of other severe psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* A Patient Health Questionnaire-9 (PHQ-9) score of ≥15 at screening
* A lifetime history of suicidal attempt
* Suicidal behavior within 30 days before screening
* Suicidal ideation corresponding to type 4 or 5 based on the Columbia-Suicide Severity
* Rating Scale (C-SSRS) within the past 30 days before screening
* Participants with confirmed diagnosis of bulimia nervosa disorder

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Disposition Index (oDI) | Baseline and 6 months
  The oDI value is the product of total responsivity index and insulin sensitivity. The change in oDI from baseline to 6M on treatment is calculated as the difference between 6M oDI value and baseline oDI value. The oDI measures the ability of beta-cell to respond to a glucose stimulus.
Change in Protein Density Fat Fraction (PDFF) | Baseline and 6 months
  The change in PDFF from baseline to 6M on treatment is calculated as the difference between 6M PDFF value and Baseline PDFF. It provides an accurate, non-invasive, reproducible, quantitative, and precise estimation of liver fat content. The expected changes in MRI-PDFF from baseline to 6M is ≥ 5.8% reduction compared to the placebo group.

SECONDARY OUTCOMES:
Change in Oral glucose tolerance test (OGTT) derived biomarkers: oDI | Baseline and 9 months
  Change in oDI from baseline to 9M after the wash-out period, calculated as the difference between 9M oDI value and baseline oDI value. This is similar to Outcome 1 except measured at 9M.
Change in OGTT derived biomarkers: fasting insulin | Baseline and 6 months
  Change in fasting insulin calculated as 1/Fasting Insulin [1/IF] from baseline to 6M.
Change in OGTT derived biomarkers: fasting insulin | Baseline and 9 months
  Change in fasting insulin calculated as 1/Fasting Insulin [1/IF] from baseline to 9M.
Change in OGTT derived biomarkers: c-peptide | Baseline and 6 months
  Change in c-peptide from baseline to 6M calculated as [change in C-peptide from 0-30min]
  /[change in glucose from 0-30 min]. This computes for early c-peptide response to oral glucose.
Change in OGTT derived biomarkers: c-peptide | Baseline and 9 months
  Change in c-peptide from baseline to 9M calculated as [change in C-peptide from 0-30min]
  /[change in glucose from 0-30 min]. This computes for early c-peptide response to oral glucose.
Change in OGTT derived biomarkers: fasting c-peptide | Baseline and 6 months
  Change in fasting c-peptide from baseline to 6M calculated as Fasting C-peptide/Fasting Insulin.
Change in OGTT derived biomarkers: fasting c-peptide | Baseline and 9 months
  Change in fasting c-peptide from baseline to 9M calculated as Fasting C-peptide/Fasting Insulin.
Time to glucose peak | Baseline
  Identification of time to glucose peak during OGTT at baseline.
Time to glucose peak | 6 months
  Identification of time to glucose peak during OGTT at 6M.
Time to glucose peak | 9 months
  Identification of time to glucose peak during OGTT at 9M.
Glucagon levels | Baseline
  Identification of glucagon levels during OGTT at baseline.
Glucagon levels | 6 months
  Identification of glucagon levels during OGTT at 6M.
Glucagon levels | 9 months
  Identification of glucagon levels during OGTT at 9M.
Incretin effect | 6 months
  Estimated as the ratio between total insulin responses during OGTT and IVGTT at the end of treatment and expressed as percentage. It is computed by: [100% × (AUCins OGTT - AUCins IVGTT)/AUCins OGTT].
Incretin effect | 9 months
  Estimated as the ratio between total insulin responses during OGTT and IVGTT at the end of the wash-out period and expressed as percentage. It is computed by: [100% × (AUCins OGTT - AUCins IVGTT)/AUCins OGTT].
Change in Protein Density Fat Fraction (PDFF) | Baseline and 9 months
  The change in PDFF from baseline to 9M after the wash-out period is calculated as the difference between 9M PDFF value and Baseline PDFF. It provides an accurate, non-invasive, reproducible, quantitative, and precise estimation of liver fat content. The expected changes in MRI-PDFF from baseline to 9M is ≥ 5.8% reduction compared to the placebo group.
Fractional rates of de Novo Lipogenesis (DNL) | Baseline
  It is the measure of contribution of hepatic DNL and plasma free fatty acid reesterification to plasma triglyceride secretion at baseline. It is calculated by F = plasma palmitate enrichment/(22 X plasma deuterium enrichment). F is the fraction of palmitate synthesized during the time between the loading dose of the deuterium-labeled water and the collection time.
Fractional rates of de Novo Lipogenesis (DNL) | 6 months
  It is the measure of contribution of hepatic DNL and plasma free fatty acid reesterification to plasma triglyceride secretion at 6M. It is calculated by F = plasma palmitate enrichment/(22 X plasma deuterium enrichment). F is the fraction of palmitate synthesized during the time between the loading dose of the deuterium-labeled water and the collection time.
Fractional rates of de Novo Lipogenesis (DNL) | 9 months
  It is the measure of contribution of hepatic DNL and plasma free fatty acid reesterification to plasma triglyceride secretion at 9M. It is calculated by F = plasma palmitate enrichment/(22 X plasma deuterium enrichment). F is the fraction of palmitate synthesized during the time between the loading dose of the deuterium-labeled water and the collection time.
Total cholesterol | 6 months
  Measure of total cholesterol in plasma taken at 6M.
Total cholesterol | 9 months
  Measure of total cholesterol in plasma taken at 9M.
LDL cholesterol | 6 months
  Measure of LDL cholesterol in plasma taken at 6M.
LDL cholesterol | 9 months
  Measure of LDL cholesterol in plasma taken at 9M.
HDL cholesterol | 6 months
  Measure of HDL cholesterol in plasma taken at 6M.
HDL cholesterol | 9 months
  Measure of LDL cholesterol in plasma taken at 9M.
Triglycerides | 6 months
  Measures of triglycerides in plasma taken at 6M.
Triglycerides | 9 months
  Measures of triglycerides in plasma taken at 9M.

OTHER OUTCOMES:
Changes in liver fibrosis | 6 months
  Changes in fibrosis of the liver as measured by the difference between MRE Stiffness during baseline and 6M.
Changes in liver fibrosis | 9 months
  Changes in fibrosis of the liver as measured by the difference between MRE Stiffness during baseline and 9M.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Pediatric Diabetes Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No